CLINICAL TRIAL: NCT00982306
Title: Brief Interventions for Heavy Alcohol Users Admitted to General Hospital
Brief Title: Brief Interventions in General Hospital (BIG)
Acronym: BIG
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Partnerships in Care (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Jean McQueen, NHS Greater Glasgow and Clyde
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: SN08OC202
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Alcoholism
Keywords: alcohol; brief interventions; counseling; harmful/hazardous alcohol drinkers
MeSH Terms: conditions — Alcoholism | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Brief intervention — 20 minute one to one counseling session

SUMMARY:
Alcohol abuse is a widespread concern internationally with a significant threat to world health. Research suggests a relationship between heavy drinking and certain clinical presentations such as injuries, physical and psychiatric illnesses and frequent sickness absence from employment. This research aims to establish whether brief interventions delivered to harmful and hazardous alcohol drinkers admitted to hospital impacts of their alcohol consumption levels on discharge from hospital.

DETAILED DESCRIPTION:
Purpose To evaluate the effectiveness of brief interventions for hazardous and harmful alcohol abusers admitted to medical and surgical wards at the Southern General Hospital

Evidence for brief interventions in general hospital Further research is required to prove the benefits of brief interventions within general hospital, based on evidence from the Cochrane systematic review 'Brief interventions for heavy alcohol users admitted to general hospital wards' (McQueen et al 2009).

Links with national and international agendas The European Health Target12 supports a reduction in harm from alcohol drugs and tobacco. By the year 2015 the adverse health effects from the consumption of addictive substances such as alcohol should be reduced by all member states (European Health for all targets 1998) The Scottish government has set HEAT (Health improvement, efficacy and governance access and treatment) target for the NHS to deliver 149,449 alcohol brief intervention cumulatively over the period of 2008/9-2010/11 (Scottish Alcohol and Drugs Workforce 2008).

Research Design This study will employ a randomised control trial design. The primary outcome measure will be grams of alcohol consumed per week, measures will be taken at baseline, six months and one year post intervention. Secondary outcomes will consist of brief intervention's impact on hospital re-admission rates, attendance at A&E and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Scores between 3-12 on FAST
* Admitted to hospital
* Speaks english

Exclusion Criteria:

* Under 18 years
* Cognitively impaired
* Medically Unfit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption in units | 6 months and one year

SECONDARY OUTCOMES:
Hospital readmissions | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Southern General Hospital, Glasgow, United Kingdom

REFERENCES:
- [Derived] McQueen JM, Ballinger C, Howe TE. Factors associated with alcohol reduction in harmful and hazardous drinkers following alcohol brief intervention in Scotland: a qualitative enquiry. BMC Health Serv Res. 2017 Mar 8;17(1):181. doi: 10.1186/s12913-017-2093-7. PMID 28270194